CLINICAL TRIAL: NCT05541822
Title: A Phase 2 Multicenter, Open-Label, Parallel Cohort Expansion Study to Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetic Profile of ABN401 in Patients With Advanced Solid Tumors Harboring c-Mesenchymal-epithelial Transition Factor (c-MET) Dysregulation
Brief Title: To Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetic Profile of ABN401 in Patients With Advanced Solid Tumors Harboring c-MET Dysregulation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abion Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABN401-003
Record Dates: First submitted 2022-09-04; First posted 2022-09-15 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumors
Keywords: c-MET
MeSH Terms: interventions — lazertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1: Vabametkib (Experimental): Subjects will receive vabametkib 800 mg, monotherapy, administered orally once daily in 21-day cycles
  Interventions: Drug: Vabametkib
- Cohort 2: Lazertinib & Vabametkib (Experimental): Part 1 (Safety Run-in): Subjects will receive lazertinib 240 mg in combination with one of three assigned dose levels of vabametkib, administered orally once daily in 21-day cycles
  Part 2 (Random Dose Optimization): A maximum of two vabametkib dose levels will be evaluated in this part. Patients will be randomized in 1:1 ratio to vabametkib dose level 1 (selected from Part 1) plus the determined dose of lazertinib or dose level 2 (selected from Part 1) plus the determined dose of lazertinib
  Part 3 (Randomized Clinical Trial): Patients will be randomized in 1:1 ratio to optimized vabametkib dose (selected from Part 2) plus lazertinib or Standard of Care (SOC) arm. SOC arm will be decided by the time of Part 3 initiation
  Interventions: Drug: Vabametkib; Drug: Lazertinib

INTERVENTIONS:
Drug: Vabametkib — Tablets
  Route of Administration: Oral
Drug: Lazertinib — Tablets
  Route of Administration: Oral
  Arms: Cohort 2: Lazertinib & Vabametkib

SUMMARY:
ABN401-003 is a Phase 2 clinical study to assess efficacy, safety, tolerability and pharmacokinetic profile of ABN401 (vabametkib) in specific populations of advance solid tumors with c-MET alterations as monotherapy.

DETAILED DESCRIPTION:
This study will start with one cohort and it will be a parallel cohort expansion study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age or designated age of majority according to the regulatory authorities, whichever is higher.
2. Eastern Cooperative Oncology Group (ECOG) performance status (PS), 0 or 1.
3. Have a life expectancy of at least 3 months.
4. Diagnosis:

   1. must have histologically or cytologically confirmed NSCLC, advanced, recurrent, or metastatic,
   2. For Cohort 1: MET exon 14 skipping suspected by local or central biomarker assessment. [local testing is accepted for eligibility; all patients will have confirmation by central laboratory, but this result is not necessary for eligibility; local molecular pathology result will suffice]. This testing can be from archival or fresh tissue sample and/or blood specimen; any sample, any test positive subjects are eligible.
   3. For Cohort 2:

      * Non-squamous histology (confirmed by histology or cytology)
      * EGFR mutation-positive including exon 19 deletions or exon 21 L858R as detected by an FDA-approved or other validated test in a CLIA certified laboratory (sites in the US) or an accredited local laboratory (sites outside of the US) in accordance with site standard of care. (Note: A copy of the test report documenting the EGFR mutation must be included in the participant records and it must be reviewed by the Medical monitor.)
      * Radiological documentation of disease progression while on continuous treatment with the 1st line 3rd generation EGFR-TKI
      * Prior objective clinical benefit defined by either partial or complete radiological response, or durable SD (SD should last > 6 months) from the 1st line 3rd generation EGFR-TKI
      * Interval between documentation of radiological progression of disease on the 1st line 3rd generation EGFR TKI and first dose of study drug should be ≤ 60 days
      * MET amplification or overexpression from tumor sample collected following progression on 1st line 3rd generation EGFR-TKI • Amplification GCN ≥ 10 indicated by FISH (confirmed centrally, slides or image from local laboratory will be confirmed by the central pathologist) or NGS (confirmed either centrally or locally) • Overexpression indicated by IHC90+ (i.e. 3+ staining in ≥ 90% tumor cells by central test, if local IHC results are available, image from local laboratory will be confirmed by central pathologist. Despite the image submission, tissue unstained slides should be sent to central laboratory for confirmation of MET amplification or overexpression.)
5. Treatment experience

   1. Cohort 1: Anti-tumor treatment naïve subject upon refusal to receive 1st line standard of care, or not tolerated to 1st line standard of care, or progressed after standard of care with no greater than 2 prior treatment regimens (neoadjuvant, adjuvant, and maintenance therapies do not qualify as separate treatment regimens).
   2. Cohort 2: Progressed on prior the 1st line 3rd generation EGFR-TKI for the treatment of advanced/metastatic NSCLC
6. At least one measurable lesion per response evaluation criteria in solid tumors (RECIST) 1.1
7. While on study treatment and for 6 months after the last dose of study treatment, a patient must:

   1. Not breast feed or be pregnant.
   2. Not donate gametes (ie, eggs or sperm) or freeze for future use for the purpose of assisted reproduction.
   3. Wear an external condom when engaging in any activity that allows for passage of ejaculate to another person.
   4. If of childbearing potential

   i. Have a negative highly sensitive (eg, beta-human chorionic gonadotropin [β-hCG]) pregnancy test at screening and within 72 hours before the first dose of study treatment, and agree to further pregnancy tests, ii. Practice at least 1 highly effective method of contraception; if oral contraceptives are used, a barrier method of contraception must also be used.

   e. If a patient's partner is of childbearing potential, the participant must use a condom and partner of the participant must also be practicing a highly effective method of contraception. A vasectomized patient must still use a condom, but the partner is not required to use contraception.
8. Resolution of prior-therapy-related AEs (including immune-related AEs but excluding alopecia) to ≤ Grade 1 per CTCAE v 5.0, and no treatment for these AEs for at least 2 weeks prior to the time of enrollment. Alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 AEs not constituting a safety risk based on investigator's judgment are acceptable.
9. Adequate organ function as indicated by laboratory values.
10. Submit tissue and blood specimens.

<!-- -->

1. Cohort 1:

   1. All patients should submit tumor tissue/block collected from fresh biopsy or have available archival formalin-fixed, paraffin-embedded tumor tissue specimen. The archival tissue must be:

      * collected after progression from most recent prior systemic anti-cancer treatment, OR
      * If an archival tissue collected after progression to the most recent systemic anti-cancer treatment is not available, tissue samples from previous lines of treatment are acceptable.

      For fresh biopsied sample, core needle biopsy is permitted. Samples from fine-needle aspiration (FNA) is not acceptable unless the result of MET exon 14 skipping from local testing is available.
   2. All patients must submit blood samples.
2. Cohort 2:

   1. All patients should submit either fresh or archival tumor slides/block collected after progression from 1st line 3rd generation EGFR TKI. The archival tissue can be permitted ONLY IF it is collected after progression from 1st line 3rd generation EGFR TKI.
   2. All patients should submit blood samples. 11. Able and willing to comply with the protocol and the restrictions and assessments therein.

Exclusion Criteria:

1. Previous severe hypersensitivity reaction to any component of study drug(s).
2. Prior therapy

   a. Previous treatment with c-MET inhibitors or hepatocyte growth factor (HGF)-targeting therapy.

   b. For Cohort 2, prior chemotherapy for advanced, recurrent, or metastatic setting.
3. Genetic analysis results:

   1. Cohort 1: Existing genetic data from the patient's tumor tissue showing known molecular alterations which would make them eligible for targeted therapies (e.g., EGFR mutations, ALK rearrangements, KRAS mutation, ROS1 translocation, BRAF mutation, RET alteration, and NTRK fusion, etc.).
   2. Cohort 2: Patients with known molecular alterations that can't benefit from study medication (e.g., EGFR mutation known to be associated with the resistance to 3rd generation EGFR TKIs, such as C797X or insertion 20, ALK rearrangements, KRAS mutation, ROS1 translocation, BRAF mutation, RET alteration, and NTRK fusion, etc.).
4. Chronic inflammatory liver condition. History or clinical evidence of any significant liver or biliary pathology including cirrhosis, infectious disease, inflammatory conditions, steatosis, or cholangitis (including ascending cholangitis, primary sclerosing cholangitis, obstruction, perforation, fistula of biliary tract, spasm of sphincter of Oddi, biliary cyst or biliary atresia).
5. Past medical history of Interstitial Lung Disease (ILD)/pneumonitis, drug-induced or radiation ILD/pneumonitis that required steroid treatment or other immune suppressive agents, or evidence of current symptomatic interstitial lung disease or unexplained pulmonary symptoms indicative of ILD such dyspnea, cough, or fever.
6. Impairment of Gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drugs (e.g., ulcerative diseases, uncontrolled nausea, uncontrolled vomiting, uncontrolled diarrhea, or malabsorption syndrome)
7. Prior organ or stem cell transplant.
8. Known active infection with human immunodeficiency virus (HIV), human T-cell leukemia virus, type (HTLV-1), hepatitis B virus (HBV), or hepatitis C virus (HCV), unless the patients fall into below categories (patients fall into one of the a, b, c category are eligible to participate)

   1. HIV

      ✓ CD4+ cells ≥ 350 cells/µL

      ✓ No history of AIDS

      ✓ No history of opportunistic infection in the past 12 months
   2. HCV

      ✓ Undetectable viral load (Participants positive for hepatitis C antibody are eligible only if polymerase chain reaction is negative for hepatitis C RNA)
   3. HBV ✓ Concurrent HBV treatment and undetectable viral load (Participants with a past or resolved hepatitis B infection defined as the presence of hepatitis B core antibody [anti-HBc] and absence of hepatitis B surface antigen are eligible)
9. Symptomatic ascites or pleural effusion, unless clinically stable for at least two weeks following treatment for these conditions (including therapeutic thoraco- or paracentesis).
10. Known active central nervous system (CNS) primary tumor or metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are clinically stable for at least 4 weeks prior to first dose of study medication(s), have no evidence of new or enlarging brain metastases and are off steroids for at least 15 days prior to first dose of study medication(s).
11. Presence or history of a malignant disease other than disease to be treated in current protocol that has been diagnosed and/or required therapy within the past 3 years. Exceptions to this exclusion include the following: completely resected basal cell and squamous cell skin cancers, indolent malignancies that currently do not require treatment, and completely resected carcinoma in situ of any type.
12. Active infection requiring therapy. However, subject with minor infections requiring oral antibiotics, (e.g., urinary tract infection, Upper respiratory tract infection, etc.) could be eligible based on investigator's judgement.
13. Use of systemic corticosteroids > 10 mg/day prednisone or equivalent within 30 days or other immunosuppressive drugs within 30 days prior to first drug administration.
14. Patients receiving treatment with medications that meet one of the following criteria and that cannot be discontinued specified period prior to the start of treatment with study drug and for the duration of the study.

    For Vabametkib (Wash-out: 1 week)

    • Strong and moderate inhibitors/inducers of P-glycoprotein

    • Strong and moderate inhibitors/inducers of CYP3A4

    • Proton pump inhibitors (PPI)

    • Potassium-competitive acid blockers For Lazertinib
    * Strong and moderate CYP3A4 inducers
    * Medications possibly prolong QT interval or induce Torsades de Pointes
15. Has received or will receive a live vaccine within 30 days prior to the first administration of study medication. Seasonal flu vaccine that does not contain live vaccine are permitted.
16. Received an investigational product (except for EGFR TKI in Cohort 2) or treated with an investigational device within 30 days prior to first study drug administration.
17. Has been receiving: radiotherapy, chemotherapy, or molecularly-targeted agents or tyrosine kinase inhibitors (except for EGFR TKI in Cohort 2) within 2 weeks (4 weeks in case of thoracic radiotherapy to lung fields) or 5 half-lives (whichever is longer) of the start of study treatment; immunotherapy/monoclonal antibodies within 3 weeks of the start of study treatment; nitrosoureas, antibody-drug conjugates, or radioactive isotopes within 6 weeks of the start of study treatment; 7-day washout is permitted for palliative radiation (i.e. limited field, ≤ 14-day course of radiotherapy) to non-CNS lesions.
18. History or clinical evidence of any surgical or medical condition which the investigator judges as likely to interfere with the results of the study or pose an additional risk in participating e.g., rapidly progressive or uncontrolled disease involving a major organ system-vascular, ophthalmologic, cardiac (clinically important abnormalities in rhythm, conduction or morphology of resting ECG, uncontrolled hypertension, uncontrolled symptomatic heart failure), pulmonary, gastrointestinal, gynecologic, hematologic, neurologic, neoplastic, renal, endocrine, autoimmune or an immunodeficiency, or clinically significant active psychiatric or abuse disorders.
19. Is a regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol).
20. Patients with a corrected QT interval (using Fridericia's correction formula) (QTcF) of > 470 msec.
21. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medications known to prolong QT interval or induce Torsades de Pointes.
22. Congestive heart failure (CHF), defined as New York Heart Association (NYHA) class III-IV or hospitalization for CHF (any NYHA class), within 6 months of randomization.
23. An active or past medical history of pericarditis, pericardial effusion that is clinically unstable, or myocarditis. Pericardial effusion considered due to the disease under study is permitted if clinically stable at Screening.
24. (for Cohort 2) Baseline LVEF either <50% or below the lower limit of normal (LLN) per institutional guidelines, as assessed by screening echocardiogram or MUGA scan.
25. (for Cohort 2) Patients who have been receiving medications with potential for QT interval prolongation will be eligible only when the wash out period was finished.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Objective response rate (ORR) according to response evaluation criteria in solid tumors (RECIST)1.1 by Blinded Independent Central Review (BICR) | Up to 12 months
  ORR is defined as the proportion of patients who experience a complete response (CR) or partial response (PR) as measured by RECIST 1.1
Cohort 2 Part 1: Incidence of DLT (Dose Limiting Toxicity) | Up to 12 months
Cohort 2 Part 2: Optimal dose of vabametkib and lazertinib combination for Part 3 based on the risk-benefit assessment considering both ORR (Objective Response Rate) and AE (Adverse Events) | Up to 12 months
Cohort 2 Part 3: ORR (Objective Response Rate) | Up to 12 months

SECONDARY OUTCOMES:
Cohorts 1 & 2: Objective response rate (ORR) measured by RECIST 1.1 by BICR | Up to 12 months
  ORR is defined as the proportion of patients who experience a CR or PR as measured by RECIST 1.1 by BICR
Cohorts 1 & 2: Duration of response (DoR) as measured by RECIST 1.1 by BICR | Up to 12 months
  DoR as measured by RECIST 1.1 by ICR and investigator will be used. DoR is defined as the time period from documentation of disease response to disease progression.
Cohorts 1 & 2: Disease advanced control rate (DCR) as measured per RECIST 1.1 by BICR | Week 12
  DCR is defined as the proportion of patients who achieve CR, PR, and stable disease (SD) as measured per RECIST 1.1 by ICR and investigator
Cohorts 1 & 2: Progression-free survival (PFS) according to RECIST 1.1 by BICR | Up to 18 months
  PFS defined as the time from first dose of vabametkib until disease progression according to RECIST 1.1 by investigator
Cohorts 1 & 2: Overall survival (OS) according to RECIST 1.1 | Up to 18 months
  OS defined as the time from first dose of study drug until death from any cause
Cohort 1: Incidence of AEs of vabametkib | Up to 12 months
  Safety and tolerability will be a comprehensive evaluation of AEs based on:
  * Incidence of AEs (including grade 3 and 4 TEAEs)
  * Vital signs measurements
  * Clinical laboratory analyses
  * ECGs
  * Physical examination findings
  * Visual examinations
  * Concomitant medications monitored throughout the study
Cohort 2: Incidence of AEs of vabametkib with lazertinib combination | Up to 12 months
  Safety and tolerability will be a comprehensive evaluation of AEs based on:
  * Incidence of AEs (including grade 3 and 4 TEAEs)
  * Vital signs measurements
  * Clinical laboratory analyses
  * ECGs (electrocardiogram)
  * ECHO (Echocardiography) or MUGA (Multiple Gated Acquisition) scans
  * Physical examination findings
  * Visual examinations
  * Concomitant medications monitored throughout the study
Cohorts 1 & 2: Intensive Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - Tmax: Time to reach maximum concentration | Cycle 1: Days 1, 2, 15, and 16 (pre-dose). Pre-dose on Day 1 from Cycle 2 Day 1 onward until disease progression (PD), or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Sparse Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - Tmax: Time to reach maximum concentration | Cycle 1: Day 1, Even cycles: Day 1 until disease progression (PD) or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Intensive Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - Cmax: Maximum concentration | Cycle 1: Days 1, 2, 15, and 16 (pre-dose). Pre-dose on Day 1 from Cycle 2 Day 1 onward until disease progression (PD), or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Sparse Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - Cmax: Maximum concentration | Cycle 1: Day 1, Even cycles: Day 1 until disease progression (PD) or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Intensive Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - Ke: apparent first-order terminal elimination rate constant | Cycle 1: Days 1, 2, 15, and 16 (pre-dose). Pre-dose on Day 1 from Cycle 2 Day 1 onward until disease progression (PD), or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Sparse Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - Ke: apparent first-order terminal elimination rate constant | Cycle 1: Day 1, Even cycles: Day 1 until disease progression (PD) or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Intensive Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - T1/2: apparent first-order terminal elimination half-life | Cycle 1: Days 1, 2, 15, and 16 (pre-dose). Pre-dose on Day 1 from Cycle 2 Day 1 onward until disease progression (PD), or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Sparse Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - T1/2: apparent first-order terminal elimination half-life | Cycle 1: Day 1, Even cycles: Day 1 until disease progression (PD) or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Intensive Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - AUC0-t: area under the concentration-time curve from time zero to the last measurable concentration | Cycle 1: Days 1, 2, 15, and 16 (pre-dose). Pre-dose on Day 1 from Cycle 2 Day 1 onward until disease progression (PD), or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Sparse Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - AUC0-t: area under the concentration-time curve from time zero to the last measurable concentration | Cycle 1: Day 1, Even cycles: Day 1 until disease progression (PD) or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Intensive Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - AUC0-12: area under the concentration-time curve from time zero to 12 hr post-dose | Cycle 1: Days 1, 2, 15, and 16 (pre-dose). Pre-dose on Day 1 from Cycle 2 Day 1 onward until disease progression (PD), or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Sparse Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - AUC0-12: area under the concentration-time curve from time zero to 12 hr post-dose | Cycle 1: Day 1, Even cycles: Day 1 until disease progression (PD) or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Intensive Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - AUC0-24: area under the concentration-time curve from time zero to 24 hr post-dose | Cycle 1: Days 1, 2, 15, and 16 (pre-dose). Pre-dose on Day 1 from Cycle 2 Day 1 onward until disease progression (PD), or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Sparse Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - AUC0-24: area under the concentration-time curve from time zero to 24 hr post-dose | Cycle 1: Day 1, Even cycles: Day 1 until disease progression (PD) or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Intensive Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - AUC0-tau: area under the plasma concentration-time curve from time zero to next dosing | Cycle 1: Days 1, 2, 15, and 16 (pre-dose). Pre-dose on Day 1 from Cycle 2 Day 1 onward until disease progression (PD), or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Sparse Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - AUC0-tau: area under the plasma concentration-time curve from time zero to next dosing | Cycle 1: Day 1, Even cycles: Day 1 until disease progression (PD) or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Intensive Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - AUC0-∞: area under the plasma concentration-time curve from time zero to infinity | Cycle 1: Days 1, 2, 15, and 16 (pre-dose). Pre-dose on Day 1 from Cycle 2 Day 1 onward until disease progression (PD), or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Sparse Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - AUC0-∞: area under the plasma concentration-time curve from time zero to infinity | Cycle 1: Day 1, Even cycles: Day 1 until disease progression (PD) or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Intensive Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - %Extrap: percentage of AUC0-∞ obtained by extrapolation | Cycle 1: Days 1, 2, 15, and 16 (pre-dose). Pre-dose on Day 1 from Cycle 2 Day 1 onward until disease progression (PD), or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Sparse Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - %Extrap: percentage of AUC0-∞ obtained by extrapolation | Cycle 1: Day 1, Even cycles: Day 1 until disease progression (PD) or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Intensive Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - Cave: average concentration over a dosage interval | Cycle 1: Days 1, 2, 15, and 16 (pre-dose). Pre-dose on Day 1 from Cycle 2 Day 1 onward until disease progression (PD), or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Sparse Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - Cave: average concentration over a dosage interval | Cycle 1: Day 1, Even cycles: Day 1 until disease progression (PD) or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Intensive Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - FLUCP: fluctuation over a dosage interval | Cycle 1: Days 1, 2, 15, and 16 (pre-dose). Pre-dose on Day 1 from Cycle 2 Day 1 onward until disease progression (PD), or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Sparse Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - FLUCP: fluctuation over a dosage interval | Cycle 1: Day 1, Even cycles: Day 1 until disease progression (PD) or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Intensive Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - R: accumulation ratio | Cycle 1: Days 1, 2, 15, and 16 (pre-dose). Pre-dose on Day 1 from Cycle 2 Day 1 onward until disease progression (PD), or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Sparse Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - R: accumulation ratio | Cycle 1: Day 1, Even cycles: Day 1 until disease progression (PD) or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Intensive Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - CL/F: apparent systemic clearance | Cycle 1: Days 1, 2, 15, and 16 (pre-dose). Pre-dose on Day 1 from Cycle 2 Day 1 onward until disease progression (PD), or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Sparse Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - CL/F: apparent systemic clearance | Cycle 1: Day 1, Even cycles: Day 1 until disease progression (PD) or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Intensive Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - Vss/F: apparent volume of distribution at steady-state | Cycle 1: Days 1, 2, 15, and 16 (pre-dose). Pre-dose on Day 1 from Cycle 2 Day 1 onward until disease progression (PD), or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Sparse Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - Vss/F: apparent volume of distribution at steady-state | Cycle 1: Day 1, Even cycles: Day 1 until disease progression (PD) or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Intensive Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - Vz/F: apparent volume of distribution | Cycle 1: Days 1, 2, 15, and 16 (pre-dose). Pre-dose on Day 1 from Cycle 2 Day 1 onward until disease progression (PD), or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Sparse Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - Vz/F: apparent volume of distribution | Cycle 1: Day 1, Even cycles: Day 1 until disease progression (PD) or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Intensive Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - Cmin: minimum concentration during dosage interval | Cycle 1: Days 1, 2, 15, and 16 (pre-dose). Pre-dose on Day 1 from Cycle 2 Day 1 onward until disease progression (PD), or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Sparse Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - Cmin: minimum concentration during dosage interval | Cycle 1: Day 1, Even cycles: Day 1 until disease progression (PD) or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Intensive Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - Ctrough: concentration of the drug just prior to administration of next dosage | Cycle 1: Days 1, 2, 15, and 16 (pre-dose). Pre-dose on Day 1 from Cycle 2 Day 1 onward until disease progression (PD), or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)
Cohorts 1 & 2: Sparse Sampling - Pharmacokinetic (PK) parameter from plasma vabametkib concentration - Ctrough: concentration of the drug just prior to administration of next dosage | Cycle 1: Day 1, Even cycles: Day 1 until disease progression (PD) or discontinuation of treatment for any other reason. Each cycle is 21 days (Up to approximately 6 years)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (4):
  - Cancer Care of North Florida, PA (Lake City Cancer Care, LLC) - Medical Oncology, Lake City, Florida
  - Mid Florida Center, Orange City, Florida
  - The Henry Ford Cancer Institute, Detroit, Michigan
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- South Korea (14):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Boramae Medical Center, Dongjak, Seoul
  - Korea University Anam Hospital, Seoul, Seoul
  - Severance Hospital, Sinchon-dong, Seoul
  - Chungbuk National University Hospital, Cheongju-si
  - Gachon University Gil Medical Center, Incheon
  - Gyeongsang National University Hospital, Jinju
  - Seoul National University Bundang Hospital, Seongnam-si
  - Kangbuk Samsung Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St Mary's Hospitals, Seoul
  - The Catholic University of Korea St Vincents Hospital, Suwon
- Taiwan (6):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Hospital, Liouying, Tainan
  - National Taiwan University Cancer Center (NTUCC), Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No